CLINICAL TRIAL: NCT03185442
Title: Evaluation of Central Cerebral Effects of Pulsed Dosed Radiofrequency (PRF) on the Lumbar Dorsal Root Ganglion (DRG) Using Functional Magnetic Resonance Imaging (fMRI).
Brief Title: Cerebral Effects of Pulsed Radiofrequency on the Lumbar Dorsal Root Ganglion With Functional Magnetic Resonance Imaging.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: fMRI-PRF-DRG v 1.0
Record Dates: First submitted 2017-05-22; First posted 2017-06-14 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Lumbar Radiculopathy; Chronic Disease
Keywords: fMRI; PRF
MeSH Terms: conditions — Radiculopathy; Chronic Disease | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRF-fMRI (Experimental)
  Interventions: Device: Pulsed Radiofrequency

INTERVENTIONS:
Device: Pulsed Radiofrequency — Pulsed Radiofrequency is performed if the sensory threshold is below 0.5 volts, the PRF consists of 380 pulses

SUMMARY:
Evaluation of central (cerebral) effects of Pulsed RadioFrequency (PRF) on the lumbar DRG (Dorsal Root Ganglion), using fMRI (functional Magnetic Resonance Imaging ). Feasibility study (after which an interim analysis is done): 5 subjects in order to detect measurable central effects inducted by PRF on DRG, follow up study 20. Total amount of subjects 25.

DETAILED DESCRIPTION:
Detect and prove the central effects of PRF and show the objective working mechanism.

PRF is often used technique to alleviate chronic radicular neuropathic pain, although good clinical results are observed the precise (central ) working mechanism is still unknown. This study aims to find the central working mechanism.

The investigator postulate the existence of central -cerebral effect of PRF on the DRG (dorsal root ganglion). If the investigator can detect the effect using fMRI and demonstrate the objective unequivocal proof that PRF on the DRG works than the investigator will be able to promote this technique for further use in the chronic pain states.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 y
* Radicular pain in lumbar region more than 6 weeks, neuropathic

Exclusion Criteria:

* Coagulopathy
* Implanted PM or SCS device
* Pregnancy
* Unwilling to undergo MRI
* Psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Central working mechanism | 6 weeks
  fMRI-BOLD

SECONDARY OUTCOMES:
Central working mechanism | 3 times in 6 weeks
  Numeric Rating Scale (NRS)
Central working mechanism | 2 times in 6 weeks
  Douleur Neuropathique Questionnaire 4 (DN 4)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier De Coster, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Patrice Forget, PhD MD, Study Director — Universitair Ziekenhuis Brussel; Jan Poelaert, PhDMD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Pain Clinic Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No